CLINICAL TRIAL: NCT05897463
Title: Breast and Nipple Neurotization Via Elongation of the Lateral Cutaneous Branches Using Intercostal Branches
Brief Title: Nipple Neurotization
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Jung-Ju Huang, Associate Professor, Chang Gung Memorial Hospital
Other Study IDs: 202201302B0
Record Dates: First submitted 2023-05-23; First posted 2023-06-09 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Breast Reconstruction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Neurotized
- Non-neurotized

SUMMARY:
A retrospective chart review will be conducted to identify patients receiving breast reconstruction and simultaneous breast neurotization. Their reconstructed breasts will be included as study group. Patients receiving breast reconstruction without neurotization will be included as negative control group. Their contralateral normal breasts in the study and the negative control group will be included as positive control. Patients' demographic data, their breast cancer treatment parameters, such as the staging, previous radiotherapy history, postmastectomy radiotherapy, neoadjuvant and adjuvant chemotherapy will be included. The reconstruction results will be evaluated as well.

Statistics Data will be analyzed using graphing and statistical analysis software. Independent t test will be applied to calculate continuous variables in demographic values, while Chi-square will be applied to calculate categorical variables such as postoperative complications. A probability of less than 0.05 will be considered significant.

Potential risks: No

Confidentiality:

All the patient identifiable information, which includes name, chart number and birthday, involved in the study will be strictly confidential.

ELIGIBILITY:
Inclusion Criteria:

* patients who received breast reconstruction and neurotization from July 2019 to August 2022 from a single breast reconstruction surgeon.
* patients who received breast reconstruction without neurotization were included as the non-neurotized group.

Exclusion Criteria:

* patients unable to complete the follow-up were excluded from the study

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients who received breast reconstruction and neurotization from July 2019 to August 2022 from a single breast reconstruction surgeon.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Changes of monofilament force at 6, 12, 18, 24, and 30 months post-operatively | post-operative 6, 12, 18, 24, and 30 months

CONTACTS AND LOCATIONS:
Locations (1):
- ChangGungMH, Taoyuan District, Taiwan